CLINICAL TRIAL: NCT00338416
Title: An Open-Labeled Pilot Study to Evaluate the Effects of High Dose PROCRIT (Epoetin Alfa) in Maintaining Hemoglobin Levels in Anemic Cancer Patients Receiving Chemotherapy on a Every Three Week Regimen
Brief Title: An Efficacy and Safety Study of PROCRIT (Epoetin Alfa) in Cancer Patients Receiving Chemotherapy Every Three Weeks
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Ortho Biotech Products, L.P. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR004612
Record Dates: First submitted 2006-06-16; First posted 2006-06-20 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-04

CONDITIONS: Cancer; Anemia
Keywords: Chemotherapy Induced Anemia; PROCRIT (Epoetin alfa); Chemotherapy; Epoetin alfa
MeSH Terms: conditions — Neoplasms; Anemia | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: Epoetin alfa

SUMMARY:
The purpose of this study is to determine the effectiveness and safety of PROCRIT (Epoetin alfa) at a starting dose of 60,000 Units (U) once every week (QW) to a target hemoglobin (Hb) of 12 g/dL (Initiation Phase), followed by a dose of 80,000 Units once every three weeks (Q3W) to maintain a Hb range of 11.5 to 12.5 g/dL (Maintenance Phase) in cancer patients receiving chemotherapy.

DETAILED DESCRIPTION:
Epoetin alfa administered three times weekly (150 U/kg) or once weekly (40,000 U) results in a response rate (defined as >= 2 g/dL Hb increase or Hb >= 12 g/dL) of approximately 65% of anemic chemotherapy patients and produces a mean hemoglobin (Hg) rise of 1.8 g/dL. Higher weekly dosing of epoetin alfa may result in a higher response rate and a more timely mean hemoglobin rise while remaining safe. Additionally, limited data are available to show whether epoetin alfa maintenance therapy can be administered less frequently than weekly and still maintain hemoglobin levels. This is an open label, multicenter, non-randomized study to determine the safety and effectiveness of epoetin alfa given to cancer patients receiving chemotherapy every three weeks.

Patients will receive injections of PROCRIT (Epoetin alfa) 60,000 Units (U) once weekly (QW) under the skin for up to 12 weeks (Initiation Phase) to achieve a hemoglobin (Hg) level of 12 g/dL until next full chemotherapy cycle. At that time they will begin the Maintenance Phase and will receive up to 4 injections of Epoetin alfa 80,000 U every 3 weeks (Q3W) under the skin for up to an additional 12 weeks. Doses will be held and adjusted downward if hemoglobin level rises to >13 g/dL or if a very rapid hemoglobin response occurs (e.g., an increase of more than 1.3 g/dL in a 2-week period).

Safety evaluations include clinical laboratory tests (hemoglobin and hematocrit), vital sign measurements (blood pressure), and adverse events. In addition, the antibodies that have developed against erythropoietin will be evaluated in patients who receive multiple doses of PROCRIT (Epoetin alfa). Patients will receive injections of Epoetin alfa 60,000 Units (U) once weekly (QW) under the skin for up to 12 weeks (Initiation Phase) to achieve a hemoglobin (Hg) level of 12 g/dL until next full chemotherapy cycle. At that time they will begin the Maintenance Phase and will receive up to 4 injections of Epoetin alfa 80,000 U every 3 weeks (Q3W) under the skin for up to an additional 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of non-myeloid malignancy and receiving chemotherapy
* Baseline Hb of <= 11 g/dL
* Planned chemotherapy for a minimum of 15 weeks to be administered every 3 weeks
* Female patients with reproductive potential must have a negative serum pregnancy test at screening.

Exclusion Criteria:

* No uncontrolled hypertension or recent history (within 6 months) of uncontrolled cardiac arrhythmias
* No pulmonary embolism
* or thrombosis
* No transfusion of white blood cells or packed red blood cells within 28 days of Epoetin alfa treatment
* No prior treatment with Epoetin alfa or any other erythropoetic agent within the previous three months

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2003-03; Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving >= 2 g/dL Hb increase from baseline or Hb >= 12 g/dL in the Initiation Phase (up to 12 weeks).

SECONDARY OUTCOMES:
Proportion of patients with >=1 g/dL Hb increase from baseline (up to 1.9 g/dL) in the Initiation Phase; those maintaining Hb level >11 g/dL (up to 11.4 g/dL); and those maintaining Hb level 11.5 to 12.5 g/dL in the Maintenance Phase (up to 12 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Montoya VP, Xie J, Williams D, Woodman RC, Wilhelm FE. An extended maintenance dosing regimen of epoetin alfa 80,000 U every 3 weeks in anemic patients with cancer receiving chemotherapy. Support Care Cancer. 2007 Dec;15(12):1385-92. doi: 10.1007/s00520-007-0263-6. Epub 2007 May 31. PMID 17541653
- See also: An Open-label Pilot Study to Evaluate the Effects of High Dose PROCRIT (Epoetin alfa) in Maintaining Hemoglobin Levels in Anemic Cancer Patients Receiving Chemotherapy on an Every 3 Week Regimen — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=606&filename=CR004612_CSR.pdf